CLINICAL TRIAL: NCT00337350
Title: A Double-Blind, Placebo-Controlled Trial of Rosiglitazone for Clozapine Induced Glucose Metabolism Impairment: Bergman's Minimal Model Analysis
Brief Title: Rosiglitazone for Clozapine Induced Glucose Metabolism Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, David C. Henderson, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 2003-P-000014
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Glucose Metabolism; Insulin Resistance
MeSH Terms: conditions — Schizophrenia; Insulin Resistance | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- rosiglitazone (Active Comparator): rosiglitazone 4mg/day
  Interventions: Drug: rosiglitazone
- placebo (Placebo Comparator): matched placebo for 4mg rosiglitazone
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rosiglitazone — Rosiglitazone 4mg, one capsule per day for eight weeks
  Arms: rosiglitazone
Drug: placebo — matched placebo for rosiglitazone 4mg/day
  Arms: placebo

SUMMARY:
We propose an eight-week, double-blind, placebo-controlled trial of rosiglitazone in schizophrenia subjects treated with clozapine using Bergman's Minimal Model (MINMOD) intravenous glucose tolerance test. Bergman's Minimal Model analysis with frequent sampled intravenous glucose tolerance test (FSIVGTT) provides a sensitive and reliable method to measure glucose effectiveness, insulin secretion and insulin sensitivity. The MINMOD determines the relationship between insulin sensitivity, insulin secretion and the degree of obesity and can be used to study drug effects upon these variables.

DETAILED DESCRIPTION:
This study is an eight-week, double-blind, placebo-controlled trial of rosiglitazone in schizophrenia subjects treated with clozapine using Bergman's Minimal Model Analysis (MINMOD) frequent sampled intravenous glucose tolerance test (FSIVGTT) for examination of glucose metabolism. Rosiglitazone, used for the treatment of type 2 diabetes, improves glycemic control by improving insulin sensitivity in target tissues while increase glucose uptake and improving signaling between insulin and glucose transporters. The MINMOD determines the relationship between insulin sensitivity, insulin secretion and the degree of obesity and can be used to study drug effects upon these variables. The computer program estimates glucose effectiveness (SG), insulin sensitivity (SI), and the acute insulin response to glucose (AIRG) from glucose and insulin values measured during the FSIVGTT.

The site for subject enrollment, clinical assessment and collection of blood samples at weeks 2, 4, and 6 will be at the Freedom Trail Clinic of the Erich Lindemann Mental Health Center. The FSIVGTT and blood samples at baseline and week 8 will be conducted at the Mallinckrodt General Clinical Research Center at Massachusetts General Hospital. Subjects will include 50 clozapine treated patients with the diagnosis of schizophrenia or schizoaffective disorder. Subjects will be matched according to baseline fasting glucose.

Subjects will be maintained on their pre-study medication. During the baseline assessment, a member of the research team will conduct the PANSS (Positive and Negative Symptom Subscale) and HAM-D (Hamilton Rating Scale for Depression) which will be repeated at weeks 4 and 8 to determine baseline and subsequent changes in psychopathology. The neuropsychological battery will be administered at baseline and week 8 and will consist of: North America Adult Reading Test, Trail Making, Degraded Stimulus Continuous Performance Test, California Verbal Learning Test, Faces and Family Picture subtests from WMS-III, Wisconsin Card Sorting Test, Letter and Category Fluency, Letter-Number Sequencing, and Grooved Peg Board. Baseline medical evaluation will include weight, height, vital signs, AIMS score, a 12-lead EKG and a physical examination.

Subjects will be instructed to eat a diet high in carbohydrates for three days before the FSIVGTT. They are instructed to fast for 12 hours preceding the test. On the morning of the test, subjects will be admitted to the General Clinical Research Center at Massachusetts General Hospital. A nutritional assessment will be performed. Baseline blood samples for fasting glucose, basic chemistry profiles, liver enzymes, complete blood count (cbc), insulin, prolactin, lipid profile, glycohemoglobin, leptin, clozapine serum levels and cortisol will be drawn. Glucose 0.3 g/kg body weight will be infused. Approximately 35 2 cc blood samples will be withdrawn for measurement of glucose and insulin concentration. At minute 20, 0.05 units/kg of insulin will be administered as an intravenous bolus injection.

Following baseline FSIVGTT, subjects will be randomized, double-blind, to either rosiglitazone or placebo. Subjects randomized to receive medication will receive rosiglitazone 4mg po qd for eight weeks or until study end. Subjects will be monitored for symptoms of diabetes at weeks 2, 4, and 8. Subjects will be evaluated at weeks 2, 4, and 8 including measurements of blood pressure, pulse and weight. Adverse events will be monitored at weeks 2, 4, and 8 with the AMDP-5, a survey of side effects and somatic symptoms. The Medical Outcomes Study Short Form-12 (SF-12) will be used to measure general health status and function. The SF-12 will be performed at baseline, weeks 4, and 8 or study end.

A cbc will be performed every two weeks, consistent with the requirements for treatment with clozapine. At week four, a fasting glucose, insulin level, and liver function tests will be performed. At the end of the eighth week, the FSIVGTT will be repeated and blood samples will be obtained for fasting glucose, basic chemistry profiles, liver enzymes, complete blood count (cbc), insulin, prolactin, lipid profile, glycohemoglobin, leptin, clozapine serum levels and cortisol. All other aspects of the subjects care will be treatment as usual.

Potential risks associated with an intravenous line include bruising at the site, bleeding and the risk of infection. During the procedure patient may experience symptoms of low blood glucose including lightheadedness, dizziness, weakness, irritability, sweating, tremor, tachycardia, anxiety, and hunger. The amount of blood drawn with each FSIVGTT is approximately 150 cc. A low risk of anemia exists secondary to the FSIVGTT; anemia has also been a side effect of treatment with rosiglitazone. Treatment with rosiglitazone has been associated with side effects including accidental injury (cuts and abrasions), headache, back pain, anemia, edema, weight gain, decreased white blood cell count, increases in total cholesterol, LDL, and HDL and decreases in free fatty acids. Phlebotomy may produce discomfort, bruising, and rarely, infection. While the clinical assessment may be stressful, the questions contained in the SCID and PANSS do not differ from those asked in routine clinical evaluations.

Potential benefits to the subject include a comprehensive diagnostic re-evaluation, screening blood tests, and estimation of risk of diabetes. The results of the tests will be shared with patients and clinicians and may contribute to medical management by helping the patient's physician in deciding if an intervention is required to reduce the risk of diabetes. An increased understanding of the process by which clozapine induces glucose intolerance and the awareness that diabetes and its complications can be prevented with concomitant treatment with an insulin sensitizer are potential benefits to this population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-65 years
* Diagnosis of schizophrenia, any subtype, schizoaffective disorder, any subtype or schizophreniform disorder
* Well established compliance with out-patient medications
* Current treatment with clozapine for a minimum of one year
* Evidence of insulin resistance: impaired fasting glucose (glucose ≥100 mg/dl) or hyperinsulinemia (fasting insulin ≥ 15 ng/dl) or a HOMA-IR (homeostasis model assessment for insulin resistance) (fasting glucose X fasting insulin/22.5) ≥2 or a SI (insulin sensitivity index)

Exclusion Criteria:

* Inability to provide informed consent
* Current substance abuse
* Significant medical illness, including congestive heart failure, severe cardiovascular disease, renal disease (serum creatinine > 1.5), anemia (Hemoglobin < 11.0 gm/dL) or psychiatrically unstable
* Severe hepatic impairment, active liver disease or increased serum transaminase levels (ALT>2.0X upper limit of normal) If at any time, ALT increases to 2X ULN, the subject's participation in the study will be terminated.
* Women of child bearing potential who are pregnant, breastfeeding, or who are unwilling or unable to use an effective form of birth control during the entire study
* Treatment with agents that induce weight loss
* History of diabetes mellitus or thyroid disease
* Current treatment with an oral hypoglycemic agent or insulin
* Known hypersensitivity to rosiglitazone or any of its components
* Fasting Glucose >126 mg/dL11. Treatment with other atypical antipsychotic agents thought to impair glucose metabolism (olanzapine) or low potency conventional agents (thioridazine, chlorpromazine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Henderson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Schizophrenia Program, Boston, Massachusetts, United States

REFERENCES:
- [Background] AMDISEN A. DRUG-PRODUCED OBESITY. EXPERIENCES WITH CHLORPROMAZINE, PERPHENAZINE AND CLOPENTHIXOL. Dan Med Bull. 1964 Oct;11:182-9. No abstract available. PMID 14209068
- [Background] Bergman RN. Lilly lecture 1989. Toward physiological understanding of glucose tolerance. Minimal-model approach. Diabetes. 1989 Dec;38(12):1512-27. doi: 10.2337/diab.38.12.1512. PMID 2684710
- [Background] Cohen S, Chiles J, MacNaughton A. Weight gain associated with clozapine. Am J Psychiatry. 1990 Apr;147(4):503-4. doi: 10.1176/ajp.147.4.503. PMID 2316740
- [Background] Cosway R, Strachan MW, Dougall A, Frier BM, Deary IJ. Cognitive function and information processing in type 2 diabetes. Diabet Med. 2001 Oct;18(10):803-10. doi: 10.1046/j.1464-5491.2001.00577.x. PMID 11678970
- [Background] Dwyer DS, Liu Y, Bradley RJ. Dopamine receptor antagonists modulate glucose uptake in rat pheochromocytoma (PC12) cells. Neurosci Lett. 1999 Oct 29;274(3):151-4. doi: 10.1016/s0304-3940(99)00712-0. PMID 10548412
- [Background] Dwyer DS, Pinkofsky HB, Liu Y, Bradley RJ. Antipsychotic drugs affect glucose uptake and the expression of glucose transporters in PC12 cells. Prog Neuropsychopharmacol Biol Psychiatry. 1999 Jan;23(1):69-80. doi: 10.1016/s0278-5846(98)00092-x. PMID 10368857
- [Background] Goldstein LE, Sporn J, Brown S, Kim H, Finkelstein J, Gaffey GK, Sachs G, Stern TA. New-onset diabetes mellitus and diabetic ketoacidosis associated with olanzapine treatment. Psychosomatics. 1999 Sep-Oct;40(5):438-43. doi: 10.1016/S0033-3182(99)71210-7. No abstract available. PMID 10479950
- [Background] Hagg S, Joelsson L, Mjorndal T, Spigset O, Oja G, Dahlqvist R. Prevalence of diabetes and impaired glucose tolerance in patients treated with clozapine compared with patients treated with conventional depot neuroleptic medications. J Clin Psychiatry. 1998 Jun;59(6):294-9. doi: 10.4088/jcp.v59n0604. PMID 9671341
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Henderson DC, Cagliero E, Gray C, Nasrallah RA, Hayden DL, Schoenfeld DA, Goff DC. Clozapine, diabetes mellitus, weight gain, and lipid abnormalities: A five-year naturalistic study. Am J Psychiatry. 2000 Jun;157(6):975-81. doi: 10.1176/appi.ajp.157.6.975. PMID 10831479
- [Background] Kay SR, Opler LA, Lindenmayer JP. Reliability and validity of the positive and negative syndrome scale for schizophrenics. Psychiatry Res. 1988 Jan;23(1):99-110. doi: 10.1016/0165-1781(88)90038-8. PMID 3363019
- [Background] Khandoudi N, Delerive P, Berrebi-Bertrand I, Buckingham RE, Staels B, Bril A. Rosiglitazone, a peroxisome proliferator-activated receptor-gamma, inhibits the Jun NH(2)-terminal kinase/activating protein 1 pathway and protects the heart from ischemia/reperfusion injury. Diabetes. 2002 May;51(5):1507-14. doi: 10.2337/diabetes.51.5.1507. PMID 11978649
- [Background] Lamberti JS, Bellnier T, Schwarzkopf SB. Weight gain among schizophrenic patients treated with clozapine. Am J Psychiatry. 1992 May;149(5):689-90. doi: 10.1176/ajp.149.5.689. PMID 1349460
- [Background] Nuechterlein KH, Dawson ME, Gitlin M, Ventura J, Goldstein MJ, Snyder KS, Yee CM, Mintz J. Developmental Processes in Schizophrenic Disorders: longitudinal studies of vulnerability and stress. Schizophr Bull. 1992;18(3):387-425. doi: 10.1093/schbul/18.3.387. PMID 1411329
- [Background] Newcomer JW, Haupt DW, Fucetola R, Melson AK, Schweiger JA, Cooper BP, Selke G. Abnormalities in glucose regulation during antipsychotic treatment of schizophrenia. Arch Gen Psychiatry. 2002 Apr;59(4):337-45. doi: 10.1001/archpsyc.59.4.337. PMID 11926934
- [Background] Saltiel AR, Olefsky JM. Thiazolidinediones in the treatment of insulin resistance and type II diabetes. Diabetes. 1996 Dec;45(12):1661-9. doi: 10.2337/diab.45.12.1661. PMID 8922349
- [Background] Segal DL, Hersen M, Van Hasselt VB. Reliability of the Structured Clinical Interview for DSM-III-R: an evaluative review. Compr Psychiatry. 1994 Jul-Aug;35(4):316-27. doi: 10.1016/0010-440x(94)90025-6. PMID 7956189
- [Background] Skre I, Onstad S, Torgersen S, Kringlen E. High interrater reliability for the Structured Clinical Interview for DSM-III-R Axis I (SCID-I). Acta Psychiatr Scand. 1991 Aug;84(2):167-73. doi: 10.1111/j.1600-0447.1991.tb03123.x. PMID 1950612
- [Background] Strachan MW, Deary IJ, Ewing FM, Frier BM. Is type II diabetes associated with an increased risk of cognitive dysfunction? A critical review of published studies. Diabetes Care. 1997 Mar;20(3):438-45. doi: 10.2337/diacare.20.3.438. PMID 9051402
- [Background] Valdes CT, Elkind-Hirsch KE. Intravenous glucose tolerance test-derived insulin sensitivity changes during the menstrual cycle. J Clin Endocrinol Metab. 1991 Mar;72(3):642-6. doi: 10.1210/jcem-72-3-642. PMID 1997519
- [Background] Ventura J, Liberman RP, Green MF, Shaner A, Mintz J. Training and quality assurance with the Structured Clinical Interview for DSM-IV (SCID-I/P). Psychiatry Res. 1998 Jun 15;79(2):163-73. doi: 10.1016/s0165-1781(98)00038-9. PMID 9705054
- [Background] Wahlin A, Nilsson E, Fastbom J. Cognitive performance in very old diabetic persons: the impact of semantic structure, preclinical dementia, and impending death. Neuropsychology. 2002 Apr;16(2):208-16. PMID 11949713
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Wirshing DA, Spellberg BJ, Erhart SM, Marder SR, Wirshing WC. Novel antipsychotics and new onset diabetes. Biol Psychiatry. 1998 Oct 15;44(8):778-83. doi: 10.1016/s0006-3223(98)00100-0. PMID 9798083

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Freedom Trial Clinic at the Erich Lindemann Mental Health Center and were studied at the Mallinckrodt General Clinical Research Center (GCRC) at Massachusetts General Hospital (MGH), Boston.
Period: Overall Study
Arm/Group | Rosiglitazone | Placebo
Started | 9 | 11
Completed | 8 | 10
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone | Placebo | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.11 (10.29) | 39.36 (7.06) | 40.15 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Insulin Sensitivity
Description: Insulin Sensitivity (IS) was assessed using a Frequently Sampled Intravenous Glucose Tolerance Test (FSIVGTT), performed at Baseline and at week 8 (study endpoint). Subjects in the Rosiglitazone treatment arm were compared to subjects in the placebo treatment arm on their change in IS between Baseline and week 8. SI was calculated from plasma glucose and serum insulin values using the MINMOD Millennium computer program. SI represents the increase in net fractional glucose clearance rate per unit change in serum insulin concentration after the intravenous glucose load (microUnits/mL).
Time Frame: baseline, week 8
Measure: Mean (Standard Deviation); unit: microUnits/mL
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 8 | 10
microUnits/mL | 3.2 (3.9) | 0.4 (0.1)
Statistical Analysis 1: Comparison: Rosiglitazone vs Placebo; Test type: Superiority or Other; p = 0.08, ANCOVA

2. Primary Outcome: Change From Baseline on Glucose Utilization (SG)
Description: Glucose utilization (SG) was assessed using a Frequently Sampled Intravenous Glucose Tolerance Test (FSIVGTT), performed at Baseline and at week 8 (study endpoint). Subjects in the Rosiglitazone treatment arm were compared to subjects in the placebo treatment arm on their change in SG between Baseline and week 8. SG was calculated from plasma glucose and serum insulin values using the MINMOD Millennium computer program. SG represents the net fractional glucose clearance rate because of the increase in glucose independent of any increase in circulating insulin concentrations above baseline.
Time Frame: baseline, week 8
Measure: Mean (Standard Deviation); unit: min^-1
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 8 | 10
min^-1 | .002 (.002) | -0.01 (0.01)
Statistical Analysis 1: Comparison: Rosiglitazone vs Placebo; Test type: Superiority or Other; p = .05, ANCOVA

3. Primary Outcome: Change From Baseline in Acute Insulin Response to Glucose (AIRG)
Description: Acute insulin response to glucose (AIRG) was assessed using a Frequently Sampled Intravenous Glucose Tolerance Test (FSIVGTT), performed at Baseline and at week 8 (study endpoint). Subjects in the Rosiglitazone treatment arm were compared to subjects in the placebo treatment arm on their change in SG between Baseline and week 8. AIRG was calculated from plasma glucose and serum insulin values using the MINMOD Millennium computer program. AIRG measures the acute(0-10 min) beta\ cell response to a glucose load calculated by the areas under the curve higher than basal insulin values. The AIRG was assessed as the incremental area under the curve (calculated by the trapezoid rule) from 0 to 10 min of the FSIVGTT.
Time Frame: baseline, week 8
Measure: Mean (Standard Deviation); unit: Units/mL per 10 minutes
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 8 | 10
Units/mL per 10 minutes | -151 (457) | 19 (22)
Statistical Analysis 1: Comparison: Rosiglitazone vs Placebo; Test type: Superiority or Other; p = 0.21, ANCOVA

ADVERSE EVENTS:
Time Frame: Baseline to week 8 (entire study)
Arm/Group | Rosiglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

LIMITATIONS AND CAVEATS:
Our findings in this study were limited by the small sample size. It is possible that with a larger sample, significant improvements might be observed not only in glucose metabolism but also in lipid metabolism.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes